CLINICAL TRIAL: NCT02995785
Title: The First Aid Skill Simulation Training of Nurses of General Wards.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 201611028RINB
Record Dates: First submitted 2016-12-12; First posted 2016-12-16 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Simulation
Keywords: Simulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental:simulation-based training (Other): Experimental
  Interventions: Other: simulation-based training; Other: traditional training
- Active comparatorr: traditional training (Other): Traditional
  Interventions: Other: traditional training

INTERVENTIONS:
Other: simulation-based training — simulation-based training:The first aid skill simulation training with discussion and debriefing(75-min) and TMS online lecture(15-min).
  Arms: Experimental:simulation-based training
Other: traditional training — traditional training:Give TMS online lecture(15-min).

SUMMARY:
[Background and Objective]First-aid skill training plays an important role in the education of nurses. How to implement stable and efficient skill is very important. (Kardong-Edgren, Oermann, Odom-Maryon, & Ha, 2010). Simulation-based workshops,or training, as the most common enhancing skills.(Topping et al., 2015) .This study was designed to assist nurses enhancing the clinical ability and safety the patients in the first aid-related skills and knowledge. The purpose of this study is to compare the two groups of(1) first aid knowledge online test. (2) first aid skills test.【Methods】This study is a general ward nurses first aid technical examination, pre-test and post-test, the random control trial. Review by the hospital ethics committee and execution date on105/12/12-107/03/08, a total of 92 cases, obtained consent of all cases, then the case will be test in our hospital clinical skills center. Subject condition: general ward nurse (minimum age> 20 years),exclusion conditions: intensive care unit nurses, emergency department nurses. Study Procedure: Subjects who obtained the informed consent were randomly assigned to the first aid skill simulation training group (FAST) or the traditional group (T) by using a computer generated number. Randomization envelopes were opened and randomization performed by the study nurse after informed consent was obtained. Each group consisted of 46 subjects. All the subjects were pre-test first aid knowledge online test, followed were pre-test first aid skills test at the Clinical Skills Center.After pre-test,the experimental group are give the first aid skill simulation training with debriefing(75-min) and online lecture(15-min).While the traditional group only give online lecture(15-min). Two weeks later, the post-test include online test and skills test for two groups. After all the data were collected by the researchers who unknown the groups, the names of the cases were removed and the scores of the two groups were compared before and after.The test Based on 2015 AHA Guidelines for CPR & ECC (2015 Adult Basic Life Support and Cardiopulmonary Resuscitation Quality & 2015American Heart Association and 2015).The data will be archived in SPSS20.0 statistical package software. Statistical methods such as T-test and Anova variance analysis are used to analyze the data【Expected Result】: The knowledge and skills in the experimental group were better than the traditional group, and the first-aid simulation skill training was helpful for the clinical emergency situations.

DETAILED DESCRIPTION:
[Background and Objective]First-aid skill training plays an important role in the education of nurses. How to implement stable and efficient skill is very important. (Kardong-Edgren, Oermann, Odom-Maryon, & Ha, 2010). Nursing first aid simulation is very often used to teaching, the teaching have significant significance of cognitive, skills, satisfaction and other indicators of achievement (Cant & Cooper, 2010),simulation-based workshops,or training, as the most common enhancing skills. (Topping et al., 2015) BLS as the basic first aid common sense and basic knowledge of resuscitation.In our hospital BLS was trained the basic knowledge and chest compression technique. According to the Department of Nursing first aid site performance check list found that the first aid equipment used unskilled , 25.5% on 2016/01 to 2016/06.The most unfamiliar techniques and knowledge of 109 nurses(all completed BLS) were as follows: 33.9% of defibrillator, 25.7% of staff role positions, 20.7% of first aid medications, and 14.7% of intubation device and LMA (Laryngeal Mask Airway ) on 105/10/1-105/10/17.This study was designed to assist nurses enhancing the clinical ability and safety the patients in the first aid-related skills and knowledge. The purpose of this study is to compare the two groups of(1) first aid knowledge online test. (2) first aid skills test.【Methods】This study is a general ward nurses first aid technical examination, pre-test and post-test, the random control trial. Review by the hospital ethics committee and execution date on105/12/12-107/03/08, a total of 92 cases, obtained consent of all cases, then the case will be test in our hospital clinical skills center. Subject condition: general ward nurse (minimum age> 20 years),exclusion conditions: intensive care unit nurses, emergency department nurses. Study Procedure: Subjects who obtained the informed consent were randomly assigned to the first aid skill simulation training group (FAST) or the traditional group (T) by using a computer generated number. Randomization envelopes were opened and randomization performed by the study nurse after informed consent was obtained. Each group consisted of 46 subjects. All the subjects were pre-test first aid knowledge online test, followed were pre-test first aid skills test at the Clinical Skills Center by eight instructors who were more than 20 years worked experience. After pre-test, the experimental group are give the first aid skill simulation training guidance on-site with discussion and debriefing(75-min) and TMS online lecture(15-min).While the traditional group only give TMS online lecture(15-min). Two weeks later, the post-test include first aid knowledge online test and first aid skills test for two groups. After all the data were collected by the researchers who unknown the groups, the names of the cases were removed and the scores of the two groups were compared before and after about(1) first aid knowledge online test. (2) first aid skills test. The test Based on 2015 AHA Guidelines for CPR & ECC (2015 Adult Basic Life Support and Cardiopulmonary Resuscitation Quality & 2015American Heart Association and 2015).First Station: Equipment testing, Second Station: Assisted with intubation and fixation, Third Station: LMA, Fourth Station: Ambu bagging, Fifth Station: Drugs, Sixth Station: Defribrator, Seventh Station: Role positioning, and Eighth Station: Leader Training. The data will be archived in SPSS20.0 statistical package software. Statistical methods such as T-test and Anova variance analysis are used to analyze the data【Expected Result】: The knowledge and skills in the experimental group were better than the traditional group, and the first-aid simulation skill training was helpful for the clinical emergency situations.

ELIGIBILITY:
Inclusion Criteria:

* general ward nurse

Exclusion Criteria:

* intensive care unit nurses, emergency department nurses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in First aid skills test at 2 Weeks. | baseline and 2 weeks.
  The test Based on 2015 AHA Guidelines for CPR & ECC (2015 Adult Basic Life Support and Cardiopulmonary Resuscitation Quality & 2015American Heart Association and 2015).The contents of the test,first station:equipment test 13%, second station:assisted with intubation and fixation 16%, third station: LMA 12%, fourth station: Ambu bagging 10%, fifth station: Drugs 12%, sixth station: Defribrator 12%, seventh station: Role positioning 17%, and eighth station: Leader Training 8%, total score is 100 points, the higher the better.

SECONDARY OUTCOMES:
Change from Baseline in First aid knowledge online test at 2 Weeks. | baseline and 2 weeks.
  The test Based on 2015 AHA Guidelines for CPR & ECC (2015 Adult Basic Life Support and Cardiopulmonary Resuscitation Quality & 2015American Heart Association and 2015). The contents of the test, 20 questions from 40 questions of random, each question 5 points, total score is 100 points, the higher the better.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing chen, Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No